CLINICAL TRIAL: NCT05728554
Title: BIC4VMR: Breakthrough Improvement Collaborative for Ventral Mesh Rectopexy
Brief Title: Breakthrough Improvement Collaborative for Ventral Mesh Rectopexy
Acronym: BIC4VMR
Status: Enrolling by invitation | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kris Vanhaecht, Professor, KU Leuven
Other Study IDs: BIC4VMR
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Learning session 1 — Learn form international report, Explain key interventions, Explain BIC methodology, Retrospective patient record analysis, Team measures
Other: Learning session 2 — Feedback report, Share (inter)national best practices, Discussion, set priorities, teaching and improvement, Retrospective patient record analysis
Other: Learning session 3 — Feedback report, Share best practices, Discussion, set priorities, teaching and improvement, Retrospective patient record analysis, Team measures

SUMMARY:
Different studies showed large variation between care processes in multiple diseases, this leads to large variation in outcomes. Better adherence to evidence-based guidelines for these diseases can reduce this variation and can improve the health outcomes.

Ventral mesh rectopexy has gained popularity in Europe to treat different rectal prolapse syndromes. This procedure has been shown to achieve acceptable anatomic results with low recurrence rates, few complications, and improvements of both constipation and fecal incontinence. However, there is limited data on the care process and outcomes. Moreover, there is no insight in the variation between different centers for patients undergoing ventral mesh rectopexy.

This study aims to map the variation in care for patients undergoing ventral mesh rectopexy in Flemish hospitals and to get an overview about the variation within and between these hospitals. Hereby, this will be a repeat of the studies for colorectal cancer, fragility hip fractures, stroke and breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years;
* Elective admission for ventral mesh rectopexy
* Total rectal prolapse
* Grade III Internal prolapse with incontinence or obstructed defaecation

Exclusion Criteria:

* Colpo posterior
* Patients diagnosed with severe dementia (DSM IV) or severe concomitant disease that may affect very short-term outcome (life expectancy less than 3 months) and hence influence deviations from standard acute care.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with rectal prolaps admitted for planned surgery
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Length of stay | through study completion, an average of 4 months
  Number of days in the hospital

SECONDARY OUTCOMES:
In-hospital complication rate | through study completion, an average of 4 months
  Re-intervention, wound complications, surgical site infection, ileus and postoperative bleeding
in-hospital mortality | through study completion, an average of 4 months
  Mortality during hospitalization
30 day readmission rate | through study completion, an average of 4 months
  Readmission rate within 30 days after discharge
30 days mortality rate | through study completion, an average of 4 months
  Mortality rate within 30 days after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium